CLINICAL TRIAL: NCT06247384
Title: The Hypotension Prediction Index in Major Abdominal Surgery - a Prospective Randomized Clinical Trial.
Brief Title: The Hypotension Prediction Index in Major Abdominal Surgery
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Jakub Szrama (Other)
Responsible Party: Sponsor-Investigator, Jakub Szrama, Principal Investigator, Poznan University of Medical Sciences
Organization: Poznan University of Medical Sciences (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: PoznanUMSHPI
Record Dates: First submitted 2024-01-09; First posted 2024-02-07 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2025-07

CONDITIONS: Hypotension During Surgery
Keywords: hypotension prediction index; major abdominal surgery; arterial pressure cardiac output; intraoperative hypotension

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- Group A - FloTrac group (No Intervention): Patients receiving standard therapy with the arterial pressure cardiac output hemodynamic monitoring
- Group B - HPI - Hypotension Prediction Index group (Experimental): Patients receiving therapy according to the hypotension prediction index hemodynamic monitoring.
  Interventions: Device: Hypotension Prediction Index Hemodynamic Monitoring

INTERVENTIONS:
Device: Hypotension Prediction Index Hemodynamic Monitoring — The application of the perioperative hemodynamic management according to the hypotension prediction index algorithm.
  Arms: Group B - HPI - Hypotension Prediction Index group

SUMMARY:
The goal of this randomized clinical trial is to compare different types of advanced hemodynamic monitoring in patients undergoing major abdominal surgery.

Participants undergoing major abdominal surgery will receive anesthesia with two different types of hemodynamic monitoring - group A will receive arterial pressure cardiac output algorithm with the FloTrac sensor and group B will receive hemodynamic monitoring with the Hypotension Prediction Index.

The main question the study aims to answer is:

• will the hypotension prediction index algorithm reduce the rate of hypotension in comparison to arterial pressure cardiac output algorithm.

DETAILED DESCRIPTION:
The fundamental aspect of the anesthetics perioperative management is to maintain hemodynamic stability, with special attention on the avoidance or reduction of the episodes of intraoperative hypotension (IOH). The incidence of intraoperative hypotension is related to an increased rate of perioperative morbidity and mortality. Even a short period of hypotension can be related to an increased risk of postoperative stroke, myocardial injury and acute kidney injury. Patients undergoing major abdominal surgery are at a high-risk of IOH because such surgeries typically require more than 2h to complete and require blood transfusion or inotrope administration. Hemodynamic monitoring and the use of goal directed therapy protocols helps to diminish the incidence of perioperative complications, however the hypotension management remains a reactive approach, an intervention is made when the hypotension has already occured. The Hypotension Prediction Index is an machine learning algorithm which allows to predict the episodes of hypotension and intervene before mean arterial pressure drops below 65 mmHg. The aim of the current study is to compare the rate of hypotension in patients undergoing major abdominal surgery with the arterial pressure cardiac output algorithm and the hypotension prediction index algorithm.

ELIGIBILITY:
Inclusion Criteria:

* Patients qualified for elective major abdominal surgery, defined as an expected duration of more than two hours, an estimated blood loss of >15% of blood volume, or an expected transfusion requirement of at least two packed red blood cells with general or combined anaesthesia.
* Patients with American Society of Anesthesiologists (ASA) status III or IV.
* Written informed consent.

Exclusion Criteria:

* Patients under 18 years
* Lack of health insurance
* Pregnancy
* Known history of congenital heart disease, severe aortic and/or mitral stenosis, heart failure and ejection fraction < 35 %
* Persistent atrial fibrillation and other arrhythmias impairing arterial pressure cardiac output monitoring

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 226 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2025-12-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Time weighed average of hypotension below 65 mmHg | "From the beginning of the anesthesia to the end of anesthesia (from induction - start of anesthesia to end of anesthesia - discharge from the post anesthesia department), assessed up to 30 days
  depth of hypotension in millimetres of mercury below a mean arterial pressure (MAP) of 65 mmHg x time in minutes spent below MAP of 65mmHg)/total duration of operation in minutes

SECONDARY OUTCOMES:
Time weighed average of hypotension below 50 mmHg | "From the beginning of the anesthesia to the end of anesthesia (from induction - start of anesthesia to end of anesthesia - discharge from the post anesthesia department), assessed up to 30 days
  depth of hypotension in millimetres of mercury below a MAP of 50 mmHg x time in minutes spent below MAP of 50 mmHg)/total duration of operation in minutes
Time weighed average of hypertension above 90 mmHg | "From the beginning of the anesthesia to the end of anesthesia (from induction - start of anesthesia to end of anesthesia - discharge from the post anesthesia department), assessed up to 30 days
  rise of hypertension in millimetres of mercury above a MAP of 90 mmHg x time in minutes spent above MAP of 90 mmHg)/total duration of operation in minutes
Time weighed average of hypertension above 100 mmHg | "From the beginning of the anesthesia to the end of anesthesia (from induction - start of anesthesia to end of anesthesia - discharge from the post anesthesia department), assessed up to 30 days
  rise of hypertension in millimetres of mercury above MAP of 100 mmHg x time in minutes spent above MAP of 100 mmHg)/total duration of operation in minutes
30 day mortality | 30 consecutive days starting from the day of the surgery
  30 day mortality
Length of hospitalisation | From the date of randomisation to the date of hospital discharge or death, whichever comes first, assessed up to 30 days
  Length of hospitalisation
Myocardial injury evaluated by postoperative troponin levels | First, second and fifth postoperative day
  Myocardial injury evaluated by postoperative troponin levels
Kidney injury evaluated by creatinine levels | First, second and fifth postoperative day
  Kidney injury evaluated by creatinine levels (increase in sCr by ≥0.3 mg/dL within 48 hours; increase in sCr to 1.5 times baseline; or urine volume less than 0.5 mL/kg/h for 6 hours)
Intraoperative fluid dose | "From the beginning of the anesthesia to the end of anesthesia (from induction - start of anesthesia to end of anesthesia - discharge from the post anesthesia department), assessed up to 30 days
  Intraoperative fluid administration
Intraoperative vasopressor dose | "From the beginning of the anesthesia to the end of anesthesia (from induction - start of anesthesia to end of anesthesia - discharge from the post anesthesia department), assessed up to 30 days
  Intraoperative vasopressor dose
Rate of intra and postoperative atrial fibrillation | "From the beginning of the anesthesia to the end of anesthesia (from induction - start of anesthesia to end of anesthesia - discharge from the post anesthesia department), assessed up to 30 days
  the occurrence of atrial fibrillation in the intraoperative and postoperative period up to 30 days

CONTACTS AND LOCATIONS:
Overall Officials: Krzysztof Kusza, Prof., Study Chair — Poznan Univeristy of Medical Sciences, Department of Anesthesiology, Intensive Therapy and Pain Management
Locations (1):
- Department of Anesthesiology, Intensive Therapy and Pain Management, Poznan, Poznań, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Szrama J, Gradys A, Nowak Z, Lohani A, Zwolinski K, Bartkowiak T, Wozniak A, Koszel T, Kusza K. The hypotension prediction index in major abdominal surgery - A prospective randomised clinical trial protocol. Contemp Clin Trials Commun. 2024 Dec 28;43:101417. doi: 10.1016/j.conctc.2024.101417. eCollection 2025 Feb. PMID 39895857